CLINICAL TRIAL: NCT03519789
Title: Cognitive and Emotional Factors in Visual Exploration Among Patients With Post-Traumatic Stress Disorder
Brief Title: Cognitive and Emotional Factors in Visual Exploration Among Patients With Post-Traumatic Stress Disorder (SAILLANCE2)
Acronym: SAILLANCE2
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_19.2; 2013-A01498-37 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Change blindness; Eye tracking; Implicit response
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-Traumatic Stress Disorders (PTSD): 30 patients with PTSD (diagnosis based on the standard DSM criteria)
- Controls: 30 healthy controls without any psychiatric or neurological diagnosis

SUMMARY:
Post-traumatic stress disorder (PTSD) is characterized by hypervigilance. In particular, previous works suggest that patients tend to scan constantly the environment for possible threats. The present project aims at investigating such attentional bias in patients with PTSD using the change blindness paradigm that offers the interesting possibility of studying sensitivity to sudden changes using ecological stimuli. More precisely, the investigators will investigate whether patients are more sensitive than matched controls to sudden changes in the visual environment and whether this hypersensitivity is specific or even stronger when visual information has an emotional content. The attentional bias will be measured using motor responses (accuracy and speed to indicate the occurrence of a change by pressing a button) as well as eye movements.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of PTSD based on the standard DSM-IV criteria,
* normal or corrected vision.
* clinically stable at the testing time

Exclusion Criteria:

* history of neurological illness or trauma that occurred in the previous six months, - pregnant and nursing women,
* drugs use in the last 24 hours,
* an acute ocular disorder.
* Participants will not be under tutorship, curatorship or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty patients with PTSD and 30 participants exposed to trauma without PTSD will be asked to detect neutral or emotional changes in 96 scenes.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Response time before the detection of neutral and emotional stimuli. | Baseline: one session
  The explicit response of the participants will be measured with the response time before the detection of neutral and emotional stimuli.

SECONDARY OUTCOMES:
Number of correct detections compared with the missed detections and false alarms. | Baseline: one session
  Performances will be measured by a sensitivity index (D prime) . This sensitivity index considers the number of correct detections compared with the missed detections and false alarms.
Total duration until the participant first fixed on a ROI. | Baseline: one session
  The implicit response will be measured by the localization and duration of fixations. All fixations outside the recording field will be excluded. The main variable will be the mean latency of the first fixation in a region of interest (ROI). This variable corresponds to the total duration until the participant first fixed on a ROI.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume VAIVA, Principal Investigator — University Hospital, Lille
Locations (1):
- University Hospital, Lille, Lille, France